CLINICAL TRIAL: NCT02359682
Title: Population Research of Sublingual Microcirculation Data of Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201409057RIN
Record Dates: First submitted 2014-11-05; First posted 2015-02-10 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Age 20-39: Patients aged from 20 to 39 years old.
  Interventions: Other: No intervention
- Age 40-59: Patients aged from 40 to 59 years old.
  Interventions: Other: No intervention
- Age 60-79: Patients aged from 60 to 79 years old.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No Intervention

SUMMARY:
This study will enrolled 90 healthy volunteers. The sublingual microcirculation will be examined by sidestreamdark-field videomicroscopy (MicroScan;Microvision Medical, Amsterdam, The Netherlands). Five video sequences (20 s) was obtained from different sublingual sites, and digitally stored the images with code numbers that did not reflect volunteers' information for later offline analysis by automated analysis software (AVA 3.0; Academic Medical Centre, University of Amsterdam, Amsterdam, The Netherlands).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged from 20 to 79 years old
* BMI ranged from 18.5 to 27 kg/m2

Exclusion Criteria:

* Systolic blood pressure > 140 mm Hg, diastolic blood pressure > 95 mm Hg, or systolic blood pressure < 90 mm Hg at enrollment
* Body temperature > 37.5 ℃ or < 35.5 ℃ at enrollment
* had been diagnose with any one of the following diseases
* hypertension
* diabetes mellitus
* peripheral arterial occlusive disease
* coronary arterial disease
* liver cirrhosis
* chronic kidney disease
* stroke
* anemia
* asthma
* chronic bronchitis
* any metabolic diseases
* any hematologic disease
* uncured cancer
* chronic uncontrolled infection
* other disease may limit daily activities
* non-native speakers

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Total small vessel density of sublingual small vessels | Once at enrollment
  Total small vessel density will be measured by Microscan and analyzed by AVA 3.0 software.

SECONDARY OUTCOMES:
Perfused small vessel density of sublingual small vessels | Once at enrollment
  Perfused small vessel density will be measured by Microscan and analyzed by AVA 3.0 software.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, anesthesiology department, Taipei, Taiwan